CLINICAL TRIAL: NCT03621800
Title: The Use of the Menthol Popsicle to Manage the Elderly Patient's Thirst in the Immediate Postoperative Period: a Randomized Clinical Trial
Brief Title: Menthol Popsicle to Manage the Elderly Patient's Thirst in the Immediate Postoperative Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Marilia Ferrari Conchon, Doctorade Student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 87689318.4.0000.5393
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Thirst
Keywords: Thirst; Elderly; Postoperative Period; Surgical Patient; Menthol; Ice; Randomized Controlled Trial

STUDY DESIGN:
Intervention Model Description: This is a study with an experimental research design. Randomized clinical trial, parallel, prospective and monocentric.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menthol popsicle (Experimental): Allocation concealment was performed through the use of individual opaque envelopes numbered externally in sequence, containing the randomly defined group information.This was performed by a researcher who did not participate in the data collection. The intensity of the initial thirst was measured by Visual Numerical Scale (VNS), which ranged from 0 (no thirst) to 10 (very intense thirst) and the discomfort of the initial thirst was measured through the Perioperative Thirst Discomfort Scale (PTDS), which is composed of 7 attributes and ranges from 0 to 14. After 20 minutes of the intervention (menthol popsicle), the final intensity and discomfort were measured using the same scales.
  Interventions: Other: Menthol popsicle
- Usual care (maintenance of fasting) (No Intervention): When allocated in the control group, the intensity of the initial thirst was measured by Visual Numerical Scale (VNS), which ranged from 0 (no thirst) to 10 (very intense thirst) and the discomfort of the initial thirst was measured through the Perioperative Thirst Discomfort Scale (PTDS), which is composed of 7 attributes and ranges from 0 to 14. After maintaining the usual care, that is, reaffirming the need for absolute fasting of food and drinks for 20 minutes, the final intensity and discomfort were measured using the same scales.

INTERVENTIONS:
Other: Menthol popsicle — The menthol popsicle composed of 0.05% menthol, 0.05% saccharin, 20ml ultrafiltered water and 2% cereal alcohol. The menthol popsicle was supported by a stick, allowing patients to taste more comfortably, with autonomy and safety
  Other Names: Menthol ice
  Arms: Menthol popsicle

SUMMARY:
Thirst is defined as the desire for water seeking and consumption, and is a prevalent symptom in the immediate postoperative period in all age groups. The elderly surgical patient, despite presenting reduced physiological responses to thirst and satiety, in clinical practice, it is observed that they have high thirst intensity. There is evidence that strategies using cold temperatures are effective in quenching thirst of the surgical patient, for this reason, the present study is justified, in order to find strategies that help to reduce thirst in this specific population that is the elderly surgical patient.

DETAILED DESCRIPTION:
The present study aims to: compare the intensity and discomfort of thirst in the use of the menthol popsicle and usual care in elderly patients in the immediate postoperative period. This is a randomized clinical trial, to be performed in a public tertiary hospital. The sample size calculation will be performed after the pilot test is conducted. Two groups will be formed through randomization. The tested intervention consists of the menthol popsicle (experimental group). Thirst intensity (primary outcome) will be measured by means of the Visual Numerical Scale and the discomfort of thirst (secondary outcome) through the Perioperative Thirst Discomfort Scale, in two moments: at the end of the first assesment of the patient and 20 minutes after the intervention. With the results of this study the intend is to offer to the scientific society subsidies on thirst presented by the elderly patients, generating evidence for the improvement of clinical practice. In addition to contributing to the preparation of health professionals in the assertive care of the elderly population, it is estimated to deepen the knowledge about appropriate and innovative interventions to manage the postoperative thirst of the elderly, considered to be this, a representative and growing part of the world population.

ELIGIBILITY:
Inclusion Criteria:

* Elective Surgeries;
* Aged 60 years and over;
* Being fasting;
* Verbalize thirst;
* Have been approved in the assesment of Safety Protocol of Thirst Management (SPTM)

Exclusion Criteria:

* Patients with ingestion and swallowing restrictions;
* Patients with self-reported allergy to mint;

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Thirst intensity | Measured at the beginning of the survey. For the experimental group, this measurement was made again 20 minutes after tasting the menthol popsicle. For the control group, this measure was made 20 minutes after the randomization
  For assesment of thirst intensity , a Visual Numeral Scale (VNS) was used, with a range from 0 (no thirst) to 10 (very intense thirst), as reported by the patients when questioned.

SECONDARY OUTCOMES:
Thirst discomfort | Measured at the beginning of the survey. For the experimental group, this measurement was made again 20 minutes after tasting the menthol popsicle. For the control group, this measure was made 20 minutes after the randomization
  The Perioperative Thirst Discomfort Scale (PTDS) was used to assess thirst discomfort. This scale is composed of 7 attributes that evaluate the signs of discomfort of perioperative thirst, as follows: dry mouth, dry lips, thick tongue, thick saliva, bad taste in the mouth, and desire to drink water. Each attribute varies between 0 (not uncomfortable), 1 (a little uncomfortable), and 2 (very uncomfortable). The final sum of the PTDS can range from 0 to 14 points, and 14 corresponds to the most intense thirst discomfort reported by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina M Galvão, Study Director — University of Sao Paulo; Ligia F Fonseca, Study Director — Universidade Estadual de Londrina
Locations (1):
- Marilia Ferrari Conchon, Cambé, PR-Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No